CLINICAL TRIAL: NCT06892990
Title: Texture and Color Enhancement Imaging (TXI) for Real-time Prediction of Histologic Changes in Patients With Inflammatory Bowel Diseases: a Comparison of White Light Endoscopy (WLE) Versus TXI
Brief Title: Texture and Color Enhancement Imaging (TXI) for Inflammation Assessment in Patients With Inflammatory Bowel Diseases
Acronym: COLORIZE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Director of the Department for Internal Medicine 1, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COLORIZE
Record Dates: First submitted 2024-09-25; First posted 2025-03-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease
Keywords: TXI; Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Intervention Model Description: This is a single-group crossover study, as the two endoscopic light modes, TXI and WLE, are alternated within the same examination in the same patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TXI mode vs. WLE mode (Experimental): Use of TXI mode vs. WLE mode for evaluating the degree of inflammation during ileocolonoscopy. Both endoscopy modes are used during the same ileocolonoscopy on the same patient. Photo documentation is taken in both modes.
  Interventions: Diagnostic Test: TXI mode vs. WLE mode

INTERVENTIONS:
Diagnostic Test: TXI mode vs. WLE mode — Experimental use of TXI mode compared to standard use of WLE to assess inflammatory activity in patients with IBD during ileocolonoscopy. Both endoscopy modes are used during the same ileocolonoscopy on the same patient.

SUMMARY:
In the context of the COLORIZE study, it is being tested whether the endoscopic light mode Texture and Color Enhancement Imaging (TXI) is non-inferior to the standard White Light Endoscopy (WLE) in assessing inflammatory activity in patients with Inflammatory Bowel Disease (IBD). For this purpose, ileocolonoscopy is performed on patients diagnosed with IBD, and standardized image documentation will be carried out in both WLE and TXI modes. Step biopsies are taken, and clinically validated, endoscopic, and histological scores are used.

DETAILED DESCRIPTION:
In order to make meaningful therapy decisions for patients with IBD, regular assessment of the extent of intestinal inflammation is necessary. This is particularly true for patients with Crohn's disease, as the inflammatory activity often does not correspond adequately to the symptoms described by the patient. Therefore, inflammatory activity is assessed not only at the time of diagnosis and during follow-up based on history, physical examination, and laboratory tests, but also through regular endoscopic examinations. The available endoscopic scores for assessing IBD were developed and validated based on the standard light setting, known as White Light Endoscopy (WLE). However, there is inadequate correlation between these scores and the most commonly used histological IBD scores. In recent years, in addition to WLE, other endoscopy modes developed for image optimization have been used for macroscopic assessment of IBD. An example of a new image-enhancing endoscopy mode is Texture and Color Enhancement Imaging (TXI; Olympus Corporation, Tokyo, Japan). The TXI mode is a directly switchable image mode on the endoscope, so it can be performed without special preparation or staining of the intestinal mucosa. Only the generated endoscopy image is digitally processed. With this endoscopy module, brightness in dark areas of an endoscopic image is selectively increased, color and surface structure are improved, making subtle tissue differences such as minor color changes more visible. There are only limited data on the use of the TXI mode for endoscopic assessment of the intestinal mucosa in patients with IBD. Only a single-center study has been conducted, which included 146 patients with ulcerative colitis, aiming to evaluate the presence of mucosal healing using WLE and TXI. In this study, the TXI mode appeared to be superior to WLE in detecting inflammatory lesions. Since an endoscopy score (so-called TXI score) that has not yet been validated in larger cohorts was used in this study, comparability between WLE and TXI has not been established. Therefore, the present project hypothesizes that predicting inflammatory activity at the histological level using the TXI mode is at least as good as using conventional WLE. Crucially, the same endoscopic score is used for both modes (TXI and WLE). Successful implementation of this research question could improve the diagnosis and monitoring of IBD patients. Moreover, if the TXI mode proves superior to WLE, it could lead to a reduction in the number of intestinal biopsies required for diagnosis, resulting in significant savings in personnel and financial resources.

The aim of the study COLORIZE is to assess the non-inferiority of TXI compared to WLE in predicting histological changes in IBD using the area under the curve (AUC) as a measure of prognostic accuracy. The hypothesis to be tested in this study is: There is no difference in the assessment of inflammatory activity in the colon and terminal ileum in chronic inflammatory bowel diseases (CED) between the TXI mode and White Light Endoscopy (WLE) when the AUC of the TXI mode (AUC_TXI) is less than the AUC of WLE (AUC_WLE) minus the non-inferiority margin δ. The null hypothesis H0 states: AUC_TXI < AUC_WLE - δ, while the alternative hypothesis H1 states that AUC_TXI ≥ AUC_WLE - δ.

A prospective, crossover study is being conducted. A total of 80 patients diagnosed with chronic inflammatory bowel disease and scheduled for outpatient ileocolonoscopy are included. After the legally required informed consent process, participating patients are asked to undertake the necessary preparation or bowel cleansing measures at home for the ileocolonoscopy.

The study consists of four parts:

Part 1: Before the start of the endoscopic examination, the patient's medical IBD therapy (current therapy and therapy of the past 12 months), current GI symptoms, and any previous GI surgeries are recorded and documented in writing using a patient questionnaire. Subsequently, an ileocolonoscopy is performed. During the withdrawal of the endoscope, the intestinal mucosa (mucosa) is assessed using the endoscopic light settings WLE and TXI. The macroscopic assessment includes the following five Regions of Interest (ROI): terminal or neo-terminal ileum, ascending colon, transverse colon, descending colon/sigmoid, rectum. One biopsy taken in all five ROI, and if necessary, additional biopsies are taken from macroscopically inflamed mucosa regardless of the ROI. Photodocumentation is performed during the examination (During the examination, at least three photos are saved per ROI, consisting of an overview photo in WLE, WLE close (close means closer to the intestinal mucosa) and TXI close). With the exception of the TXI photos, this corresponds to the standard procedure of "step biopsies" in IBD.

Part 2: Endoscopic scores (MES for ulcerative colitis, SES-CD for Crohn's disease) are determined for WLE and separately for TXI based on the photodocumentation taken during the ileocolonoscopy. Endoscopic scoring based on WLE is done by unblinded assessor 1 immediately after the examination. After completion of all ileocolonoscopies (n = 80), the entire stored image material (WLE and TXI) is re-evaluated by seven examiners, three of whom had performed a part of the ileocolonoscopies. The inflammatory activity should be assessed per photo on a scale of "inactive, mild, moderate and severe". The endoscopy photos are presented free of patient data and in random order to avoid recognition of the examinations performed by the examiners themselves.

Part 3: Pathologists at the University Hospital Ulm determine histological scores based on the collected intestinal biopsies (Geboes for ulcerative colitis, GHAS for Crohn's disease).

Part 4: The prognostic quality of TXI vs. WLE is tested using ROC curves, initially binary (inflammation vs. no inflammation). In secondary analyses, the degree of inflammation is also taken into account according to the scores obtained. The histological score is used as the gold standard.

Extended patient follow-up beyond the ileocolonoscopy procedure with biopsy collection is not necessary beyond the standard follow-up for a routine ileocolonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed inflammatory bowel disease (ulcerative colitis or Crohn's disease)
* Age ≥ 18 years

Exclusion Criteria:

* Post (procto-) colectomy
* Endoscopically impassable stenosis in the left hemi-colon
* ASA status > 2 points
* BBPS < 6 points (or < 2 points per segment)
* Severe coagulation disorder
* Pregnancy, lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of the TXI mode in assessing the degree of inflammation in the correlation between endoscopic and histological scores. | up to 12 months
  Non-inferiority of the TXI mode compared to WLE assessing inflammation in the terminal ileum or neo-terminal ileum as well as in the colon is evaluated via endoscopic and histologic scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Ulm University Hospital, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No